CLINICAL TRIAL: NCT02290470
Title: Olanzapine for the Prevention of Delayed Nausea and Vomiting in Patients With Gynecologic Cancers Receiving Carboplatin and Paclitaxel-based Chemotherapy and Guideline-directed Prophylactic Anti-emetics
Brief Title: Olanzapine Against Delayed Nausea and Vomiting in Women Receiving Carboplatin Plus Paclitaxel
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione IRCCS Istituto Nazionale dei Tumori, Milano (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Gineolanzapina
Record Dates: First submitted 2014-05-22; First posted 2014-11-14 (Estimated); Last update posted 2014-11-14 (Estimated); Status verified 2014-11

CONDITIONS: Nausea; Vomiting
Keywords: Nausea; Vomiting
MeSH Terms: conditions — Nausea; Vomiting | interventions — Olanzapine; Palonosetron; Dexamethasone; Carboplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- olanzapine Days 1-3 (Experimental): Olanzapine + Chemotherapy + Antiemetic treatment
  Patients will receive the chemotherapy drugs carboplatin and paclitaxel as well as the following anti-nausea/vomiting drugs:
  * Palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone (16 mg intravenously on the day of chemotherapy), plus
  * Olanzapine (10 mg orally on the day of chemotherapy and 10 mg orally on days 2, 3 post chemotherapy)
  Interventions: Drug: Olanzapine; Drug: Palonosetron, Dexamethasone, Carboplatin, Paclitaxel, Olanzapine
- olanzapine+Dexamethasone d 1-3 (Experimental): Olanzapine + Chemotherapy + Antiemetic treatment
  Patients will receive the chemotherapy drugs carboplatin and paclitaxel as well as the following anti-nausea/vomiting drugs:
  * Palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone (16 mg intravenously on the day of chemotherapy and 4 mg orally days 2, 3 post chemotherapy), plus
  * Olanzapine (10 mg orally on the day of chemotherapy and 10 mg orally on days 2, 3 post chemotherapy)
  Interventions: Drug: Olanzapine; Drug: Palonosetron, Dexamethasone, Carboplatin, Paclitaxel, Olanzapine
- dexamethasone days 1-3 (Active Comparator): Dexamethasone + Chemotherapy + Antiemetic treatment
  Patients will receive the chemotherapy drugs carboplatin and paclitaxel as well as usual anti-nausea/vomiting drugs:
  * Palonosetron (0.25 mg intravenously) on the day of chemotherapy, plus
  * Dexamethasone 16 mg intravenously on the day of chemotherapy (day 1), plus
  * Dexamethasone 8 mg orally on days 2 and 3 post chemotherapy
  Interventions: Drug: Olanzapine; Drug: Palonosetron, Dexamethasone, Carboplatin, Paclitaxel, Olanzapine

INTERVENTIONS:
Drug: Olanzapine — * Drug: Olanzapine 10 mg oral
  * Drug: Chemotherapy (carboplatin and paclitaxel). Patients will receive carboplatin and paclitaxel.
  * Drug: Anti-emetic treatment (palonosetron; plus dexamethasone). Palonosetron (0.25 mg IV) on the day of chemotherapy plus dexamethasone (16 mg IV on the day of chemotherapy and 8 or 4 mg (depending on the experimental arm) oral on days 2 and 3 post-chemotherapy).
  Other Names: Palonosetron; Dexamethasone; Carboplatin; Paclitaxel
Drug: Palonosetron, Dexamethasone, Carboplatin, Paclitaxel, Olanzapine — all patients enrolled in the study will receive Palonosetron, Dexamethasone, Carboplatin, Paclitaxel and olanzapine On day 1

SUMMARY:
This randomized, pilot study explores the activity of olanzapine with or without delayed dexamethasone for the prevention of delayed nausea and vomiting in women with gynecologic cancer receiving the combination of carboplatin and paclitaxel. Women treated with this regimen are particularly susceptible to chemotherapy-induced nausea and vomiting. Given anti-emetic prophylaxis with olanzapine may increase the control of delayed symptoms in women receiving carboplatin and paclitaxel.

DETAILED DESCRIPTION:
The purpose of this study is to assess if the use of olanzapine can improve control of delayed nausea and vomiting in women receiving the combination of carboplatin and paclitaxel for a gynaecologic cancer. Patients are randomized to one of three treatment arms. Please see the "Arms and Intervention" sections for more detailed information. The primary objective is to determine in each treatment group the proportion of patients achieving Complete Protection (CP; no vomiting, no rescue anti-emetics, and no more than mild nausea) during the delayed phase (days 2-5 post-chemotherapy) in the first chemotherapy cycle. The secondary objectives are:

1. To determine the proportion of patients achieving Complete Response (CR; no vomiting, and no rescue anti-emetics) during the acute (day 1 post-chemotherapy), delayed, and overall (days 1-5 post-chemotherapy) periods.
2. To determine the incidences of potential toxicities ascribed to olanzapine.
3. To assess the impact of nausea and vomiting on daily life activities in each treatment group.

Protocol treatment is to begin ≤14 days of registration. Patients will receive treatment on Days 1-3. Patients will be permitted to take rescue therapy of the treating investigator's choice based on the clinical circumstances. After completing treatment, patients will be monitored for side effects.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically documented gynaecologic cancer
* Patients who are chemotherapy naive and scheduled to receive 1-day moderately emetogenic chemotherapy (carboplatin Area under Curve (AUC) 5 plus paclitaxel).
* Women, 18 years and older
* Eastern Cooperative Oncology Group (ECOG) Performance Status of 0-2
* Adequate organ system function, defined as follows:

bone marrow: absolute neutrophil count >=1,500/L, platelets >=100,000/L liver: bilirubin 1.5 x upper limit of normal (ULN); transaminases <=2.5 x ULN kidney: creatinine <=1.5 x ULN

• Able to take oral medications

Exclusion Criteria:

* psychiatric illness or social situation that would preclude study compliance
* history of central nervous system (e.g., brain metastases, seizure disorder)
* Positive pregnancy test just before registration.
* treatment with any anti-emetic medication from 24 hours to 5 days after treatment.
* treatment with another antipsychotic agent such as risperidone, quetiapine, clozapine, phenothiazine, or butyrophenone for 30 days before or during protocol therapy.
* concurrent abdominal radiation therapy.
* concurrent quinolone antibiotic therapy.
* known hypersensitivity to olanzapine.
* vomiting and/or significant nausea (>= Common Toxicity Criteria for Adverse Events (CTCAE) grade 2) within the 24 hours before beginning chemotherapy.
* another organic cause for nausea or vomiting unrelated to chemotherapy administration.
* chronic alcoholism (as determined by the investigator).
* known cardiac arrhythmia, uncontrolled congestive heart failure or acute myocardial infarction within the previous 6 months.
* history of uncontrolled diabetes mellitus.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 81 (Estimated)
Dates: Start 2014-04; Primary Completion 2015-11 (Estimated); Study Completion 2015-11 (Estimated)

PRIMARY OUTCOMES:
Complete Protection | days 2-5 post-chemotherapy
  Proportion of patients achieving delayed Complete Protection, defined as no vomiting, no rescue anti-emetics, and no more than mild nausea measured by the Nausea and Vomiting Daily Diary/Questionnaire.

SECONDARY OUTCOMES:
Nausea scores | up to 5 days
  • Nausea scores measured by the Nausea and Vomiting Daily Diary/Questionnaire.

OTHER OUTCOMES:
Proportion of patients achieving Complete Response | up to 5 days
  • Proportion of patients achieving Complete Response, defined as no emetic episodes and no use of rescue anti-emetics measured by the Nausea and Vomiting Daily Diary/Questionnaire.
Impact of nausea and vomiting on daily life activities | day 1 (pre-chemotherapy) and day 6 (post-chemotherapy)
  • Impact of nausea and vomiting on daily life activities as measured by the Functional Living Index-Emesis Questionnaire.
Incidence of potential toxicities related to olanzapine | up to 5 days
  • Incidence of potential toxicities related to olanzapine as measured by the Nausea and Vomiting Daily Diary/Questionnaire. [Time frame: ] [Designated as safety issue: Yes]
Frequency of rescue anti-emetics | up to 5 days
  • Frequency of rescue anti-emetics measured by the Nausea and Vomiting Daily Diary/Questionnaire.

CONTACTS AND LOCATIONS:
Overall Officials: Luigi Celio, MD, Study Chair — Istituto tumori; Domenica Lorusso, MD, Principal Investigator — Istituto tumori; Gabriella Saibene, PharmD, Principal Investigator — Istituto Tumori
Locations (1):
- Istituto Nazionale dei Tumori, Milan, Milan, Italy